CLINICAL TRIAL: NCT06341179
Title: A Randomized Controlled Trial of Sleep Extension to Regulate Body Weight and Improve Learning in School-aged Children
Brief Title: Effect of Sleep Extension on Body Weight and Learning in Children (More2Sleep)
Acronym: More2Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Novo Nordisk Foundation (NNF) (Unknown); Faculty of Health, Medicine and Life Sciences, Maastricht University (Unknown); Center for Obesity Research & Education, Temple University (Unknown); Danish Research Centre for Magnetic Resonance (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2S; H-23063352 (Other: Vek.dk)
Record Dates: First submitted 2023-08-10; First posted 2024-04-02 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-01

CONDITIONS: Sleep Duration; Child Obesity; Child Development; Child Behavior
Keywords: Sleep duration; Sleep quality; Overweight and Obesity; Energy Intake; Child Development and Behavior; Well-being; Cognitive Function; Learning Ability; Memory
MeSH Terms: conditions — Pediatric Obesity; Child Behavior; Sleep Initiation and Maintenance Disorders; Overweight; Obesity; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep extension (Experimental): The sleep extension group (n=71) will receive a behavioral intervention focusing on parents putting their children to bed earlier by 60-90 minutes. Parents will be instructed only to alter their children's daily sleeping routine, and not to directly alter their diet and physical activity habits. Children and their parents will receive a behavioral intervention consisting of 6 sessions, including both in-person and virtual sessions, which will be scheduled based on the family's availability and to accommodate practicalities.
  Interventions: Behavioral: Sleep extension
- Control (No Intervention): The control group (n=71) will follow their habitual sleeping schedule. Parents will be instructed not to alter their children's daily sleeping routine, or their diet and physical activity habits. The same number and frequency of meetings (in-person or virtual) and methods of registration of bedtime/wake-up times will be used as in the sleep extension group. These meetings will be educational in nature and focus on general well-being and informing the families about the home registrations of e.g., sleep and dietary intake.

INTERVENTIONS:
Behavioral: Sleep extension — The sleep extension group will receive a behavioral intervention focusing on parents putting their children to bed earlier by 60-90 minutes. Previous studies have found this change in daily sleeping routine to be feasible and to result in 40-45 min more actual sleep. Children and their parents will receive a behavioral intervention consisting of 6 sessions, including both in-person and virtual sessions, which will be scheduled based on the family's availability and to accommodate practicalities, e.g., potential sickness or cancellations. The first two sessions will occur at the beginning of the study. These initial sessions will focus on effective behavioral strategies to enhance sleep time, including goal setting (e.g., bedtimes and wake-up times), problem-solving and preplanning, stimulus control (i.e., sleep hygiene recommendations), and positive reinforcement. Subsequent sessions will be planned with the families to occur regularly during the 12-week intervention.
  Arms: Sleep extension

SUMMARY:
More2Sleep is a randomized, controlled, parallel trial with two groups (sleep extension vs control) including 142 school-aged children (6-12 years) who have a BMI above average, defined as age- and sex-specific BMI Z-score above zero using WHO reference standards, and habitually sleep for ≤ 9 h/night. Data will be collected before and after a 3-month sleep extension intervention, and after a 6-month follow-up (at months 0, 3, and 9). The collection of data is mainly related to the main study. However, some optional examinations will be conducted on a first come, first serve basis, consisting of substudy-I (metabolic mechanisms, n=60) and substudy-II (learning mechanisms, n=142).

The primary objective is to assess the effects of sleep extension by ~45 min/night, achieved by going to bed 60-90 min earlier, on adiposity and learning ability in school-aged children who have a BMI for age and sex above average, and sleep less than recommended for their age.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-12 years old (inclusive range).
* Weight status: having a BMI above average, defined as an age- and sex-specific BMI Z-score above zero using reference standards from the WHO.
* Sleep duration: sleeping ≤9 h/night on the basis of sleep diaries filled in by the children's parents, based on recommendations by the American Academy of Sleep Medicine and the Sleep Health Foundation.

Exclusion Criteria:

* Any genetic, neurological, endocrinological or psychiatric condition that affects growth, metabolism, eating behaviors, cognitive function, or body weight (for example: dwarfism, epilepsy, attention deficit hyperactivity disorder, head trauma, β-thalassemia, hypothyroid-ism, hyperthyroidism, type I diabetes).
* Any sleep-related disorder (for example: obstructive sleep apnea, parasomnias, narcolepsy, restless leg syndrome).
* Regular use of prescribed or over-the-counter medications that influence study outcomes.
* Irregular school schedule.
* If a child's parents live separately, the child is allowed to sleep at both households. How-ever, if one of the parents does not wish to carry out the sleep intervention and follow given instructions, then the child should only sleep at their household Friday, Saturday and/or Sunday night.
* In the circumstance where the child does not speak or understand Danish, the child's parents do not have to speak or understand Danish, as long as both parties can speak and understand English.
* Participation in other research studies.
* Metal implants and claustrophobia (only for substudy-II).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 142 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
BMI Z-score | Assessed at months 0, 3 and 9
  BMI (in kg/m^2) will be calculated from weight and height (secondary outcomes), and the age- and sex-specific BMI Z-score (in units of standard deviation from the reference population mean) will be computed using international (WHO) data
Learning ability: skill learning | Assessed at months 0 and 3
  Skill learning ability will be measured as motor memory assessed as 24h retention after skill practice - I.e. total within and between session effect (range: from "low" = 0 to "high" = 100, unitless)
Learning ability: Explicit memory | Assessed at months 0 and 3
  Explicit memory assessed as 24h retention after word list memory encoding - I.e. total within and between session effect. Number of correctly recalled words in a 2-minute standardized task (range: from 0 to 20)

SECONDARY OUTCOMES:
Body fat percent | Assessed at months 0, 3 and 9
  Body fat in % of total body mass (total fat mass divided by total body weight) will be measured by a whole-body dual-energy X-ray absorptiometry (DXA) scan
Total fat mass (FM) | Assessed at months 0, 3 and 9
  Body FM (in grams) will be measured by a whole-body dual-energy X-ray absorptiometry (DXA) scan
Total lean mass (LM) | Assessed at months 0, 3 and 9
  Body LM (in grams) will be measured by a whole-body dual-energy X-ray absorptiometry (DXA) scan
Bone mineral content (BMC) | Assessed at months 0, 3 and 9
  BMC (in grams) will be measured by a whole-body dual-energy X-ray absorptiometry (DXA) scan
Bone mineral density (BMD) | Assessed at months 0, 3 and 9
  Areal BMD (in grams/cm^2) will be measured by a whole-body dual-energy X-ray absorptiometry (DXA) scan
Dietary energy intake | Assessed at months 0, 3 and 9
  Daily energy intake (in kcal/day) will be assessed with a three-day 24-hour recall interview on www.myfood24.org (daily averages will be computed)
Dietary protein, carbohydrate, fiber, and fat intakes | Assessed at months 0, 3 and 9
  Macronutrient intakes (in grams/day) will be assessed with a three-day 24-hour recall interview on www.myfood24.org (daily averages will be computed)
Subjective hunger | Assessed at months 0 and 3
  Subjective level of hunger (range: from "very hungry" = 1 to "not hungry at all" = 5) in the fasting state and at 1 and 2 hours after a standardized breakfast will be measured by using an image-based visual analog scale (VAS)
Physical activity (PA) time: total PA and MVPA | Assessed at months 0, 1.5,3 and 9
  The time (in min/day) spent being physically active regardless of intensity (total PA) and the time (in min/day) spent on moderate-to-vigorous-physical-activities (MVPA) will be measured for 7 consecutive days (daily averages will be computed) using a wrist-worn triaxial accelerometer
Resting metabolic rate (RMR) | Assessed at months 0 and 3
  RMR (in kcal/day) will be measured with indirect calorimetry (canopy mode) the morning after an overnight fast (at least 8 hours)
Thermic effect of food (TEF) | Assessed at months 0 and 3
  TEF (in kcal) will be computed as the incremental area under the curve (above RMR) for postprandial energy expenditure (measured by indirect calorimetry) for 2 hours after consuming a standardized breakfast
Weight | Assessed at months 0, 3 and 9
  Body mass (in kg) will be measured on a digital scale to the nearest 0.1 kg
Height | Assessed at months 0, 3 and 9
  Stature (in cm) will be measured using a wall-mounted stadiometer to the nearest 0.1 cm
Total energy expenditure (TEE) | Assessed at months 0 and 3
  TEE (in kcal/day) will be measured by using the doubly labelled water method (8 urine samples over 2 weeks)
Cognitive functions: Sustained attention | Assessed at months 0, 3 and 9
  Performance in neuropsychological assessment of sustained attention ability assessed as errors during a sustained test procedure, CANTAB test battery.
Cognitive functions: Spatial working memory | Assessed at months 0, 3 and 9
  Performance in neuropsychological assessment of spatial working memory assessed as errors and strategy during the test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
Cognitive functions: Inhibitory control | Assessed at months 0, 3 and 9
  Performance in neuropsychological assessment of inhibitory control assessed as errors during the test procedure (Modified Eriksen Flanker test, Psychology Software Tools, US) and Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK)
Cognitive functions: Cognitive flexibility | Assessed at months 0, 3 and 9
  Performance in neuropsychological assessment of cognitive flexibility assessed as errors during the test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK)
School performance: mathematics performance | Assessed at months 0, 3 and 9
  Mathematics proficiency will be measured by Hogrefe math test
School performance: reading comprehension | Assessed at months 0, 3 and 9
  Danish reading proficiency will be measured by Hogrefe reading comprehension test
Neurophysiological Measurement 1 - ERP Amplitude | Assessed at months 0 and 3
  EEG activity measured as the event-related potential (ERP) amplitude during the modified Eriksen Flanker Test
Neurophysiological Measurement 2 - Cortical activity during skill learning | Assessed at months 0 and 3
  Cortical activity during skill learning will be measured as EEG power
Neurophysiological Measurement 3 - Muscle activity during skill learning | Assessed at months 0 and 3
  Muscle activity during skill learning will be measured as electromyography amplitude
Neurophysiological Measurement 4 - corticocortical functional connectivity | Assessed at months 0 and 3
  Corticocortical functional connectivity will be measured as functional coupling in EEG (scale 0-1)
Neurophysiological Measurement 5 - corticomuscular connectivity | Assessed at months 0 and 3
  Corticomuscular connectivity will be measured as functional coupling between EEG and EMG during skill learning (0-1)
Eating window | Assessed at months 0, 3 and 9.
  The parents will be asked to note on a checklist when their children start and finish eating on each registration day to estimate the duration of the daily eating window.

OTHER OUTCOMES:
Health-related quality of life: child-reported | Assessed at months 0, 3 and 9
  The total summary score of health-related quality of life (from 50 to 250), and sub-scale scores (from 10 to 50) of physical well-being, psychological well-being, autonomy and parent relation, peers and social support, and school environment, will be assessed by KIDSCREEN 27 questionnaire
Health-related quality of life: parent-reported | Assessed at months 0, 3 and 9
  The Health Related Quality of Life score (from 0 to 100), Physical Health Summary score (from 0 to 100) and Psychosocial Health summary score (from 0 to 100) will be assessed by the Pediatric Quality of Life inventory (PedsQL)-Parent report (separate version for 6-7 y and 8-9 years olds)
Mental health: parent-reported | Assessed at months 0, 3 and 9
  The total difficulties score (from 0 to 40) of the Strengths and Difficulties Questionnaire, as well as sub-scale scores (from 0 to 10) of emotional symptoms, conduct problems, hyperactivity/inattention, relationship problems and prosocial behavior
Parental Stress Scale: parent-reported | Assessed at months 0, 3 and 9
  Perceived parental stress (from 18 to 90) will be assessed by the Parental Stress Scale questionnaire
Perceived Stress Scale: child-reported | Assessed at months 0, 3 and 9
  Perceived child stress score (from 1 to 39) will be assessed by the PSS-C questionnaire
Demographics: income | Assessed at month 0
  Income level (stepwise increasing from level 1 to 7) will be reported by the parents on a demographics questionnaire
Demographics: education | Assessed at month 0
  Education level (stepwise increasing from level 1 to 8) will be reported by the parents on a demographics questionnaire
Wakefulness | Assessed at months 0, 3 and 9
  Wakefulness (score from "very awake" = 1 to "sleeping" = 8) assessed by Standford Sleepiness Scale
Handedness | Assessed at month 0
  Handedness preference (right or left) will be assessed by asking the children "Which hand do you use to write and draw?" do to determine dominant hand
Fine Motor Control | Assessed at months 0, 3 and 9
  Fine motor control will be assessed by the pegboard test (score in number of pins placed correctly)
Muscle strength | Assessed at months 0, 3 and 9
  Muscular strength of the handgrip will be measured by a handgrip dynamometer (in Newton)
Brain myelination | Assessed at months 0 and 3
  Indices of myelination in grey and white matter are estimated using R1 obtained from an MP2RAGE MRI-sequence
Brain structural connectivity and microstructure | Assessed at months 0 and 3
  Grey and white matter microstructure will be examined using diffusion-weighted imaging
Brain functional connectivity | Assessed at months 0 and 3
  Functional connectivity will be measured using resting-state function MRI (fMRI)
Vital signs: blood pressure | Assessed at months 0, 3 and 9
  Systolic and diastolic blood pressure (in mmHg) will be measured at rest by using a automatic sphygmomanometer
Cognitive functions: processing speed | Assessed at months 0, 3 and 9
  Performance in neuropsychological assessment of processing speed as choice reaction time, CANTAB test battery.
Fasting and postprandial interleukin 6 concentration | Assessed at months 0 and 3
  The concentration of IL6 (in ng/L) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Fasting and postprandial cholecystokinin concentration | Assessed at months 0 and 3
  The concentration of CKK (in pg/mL) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Fasting and postprandial peptide YY concentration | Assessed at months 0 and 3
  The concentration of PYY (in pg/mL) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Fasting and postprandial glucagon like peptide 1 concentration | Assessed at months 0 and 3
  The concentration of GLP1 (in pg/mL) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Fasting and postprandial leptin concentration | Assessed at months 0 and 3
  The concentration of leptin (in ng/mL) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Fasting and postprandial ghrelin concentration | Assessed at months 0 and 3
  The concentration of ghrelin (in pg/mL) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Fasting and postprandial tumor necrosis factor alpha concentration | Assessed at months 0 and 3
  The concentration of TNFa (in ng/L) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Fasting and postprandial C-reactive protein concentration | Assessed at months 0 and 3
  The concentration of CRP (in mg/L) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Fasting and postprandial triglyceride concentration | Assessed at months 0 and 3
  The concentration of triglyceride (in mmol/L) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Fasting and postprandial total, HDL and LDL cholesterol concentrations | Assessed at months 0 and 3
  The concentrations of total, HDL and LDL cholesterol (in mmol/L) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Fasting and postprandial insulin concentration | Assessed at months 0 and 3
  The concentration of insulin (in pmol/L) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Fasting and postprandial glucose concentration | Assessed at months 0 and 3
  The concentration of glucose (in mmol/L) will be measured in blood during fasting and at 2 hours after consuming a standardized breakfast
Vital signs: heart rate | Assessed at months 0, 3 and 9
  Heart rate (in beats per minute, bpm) will be measured at rest by using an automatic sphygmomanometer
Vital signs: temperature | Assessed at months 0, 3 and 9
  Body (skin) temperature (in degrees Celsius) will be measured telemetrically in the ear
Sleep quality: self-reported sleep duration | Assessed at months 0, 3 and 9
  Sleep duration (hour/night) will be measured by the Scandinavian Sleep Questionnaire (Child and parent-reported).
Sleep quality: self-reported latency | Assessed at months 0, 3 and 9
  Latency (minutes) will be measured by the Scandinavian Sleep Questionnaire (Child and parent-reported)
Sleep quality: self-reported awakenings | Assessed at months 0, 3 and 9
  Awakenings (number/night) will be measured by the Scandinavian Sleep Questionnaire (Child and parent-reported).
Sleep quality: self-reported tiredness/sleepiness | Assessed at months 0, 3 and 9
  Tiredness/sleepiness during the day (yes/no) will be measured by the Scandinavian Sleep Questionnaire (Child and parent-reported).
Sleep quality and architecture: Sleep stages | Assessed at months 0 and 3
  Sleep stages (distribution of sleep stages in minutes and percentages of total sleep time) will be measured by polysomnography through a one night sleep period.
Sleep quality and architecture: sleep duration | Assessed at months 0 and 3
  Total sleep time (minutes) will be measured by polysomnography through a one night sleep period.
Sleep quality and architecture: sleep latency | Assessed at months 0 and 3
  Sleep latency (minutes) will be measured by polysomnography through a one night sleep period.
Sleep quality and architecture: awakenings | Assessed at months 0 and 3
  Awakenings (number) will be measured by polysomnography through a one night sleep period.
Sleep quality and architecture: arousals | Assessed at months 0 and 3
  Arousals (number per hour) will be measured by polysomnography through a one night sleep period.
Sleep: duration | Assessed at months 0, 1.5,3 and 9
  Sleep duration (in minutes per night) will be measured by using a wrist-worn triaxial accelerometer for 7 consecutive days (the average will be computed).
Sleep: movements | Assessed at months 0, 1.5,3 and 9
  Movements (number) will be measured by using a wrist-worn triaxial accelerometer for 7 consecutive days (the average will be computed).
Sleep: awakenings | Assessed at months 0, 1.5,3 and 9
  Awakenings (number) will be measured by using a wrist-worn triaxial accelerometer for 7 consecutive days (the average will be computed).
Brain structure: cortical thickness | Assessed at months 0 and 3
  Cortical thickness (mm) will be measured by a T1-weighted MR-image (MP2RAGE).
Brain structure: volume | Assessed at months 0 and 3
  Volume (mm3) will be measured by a T1-weighted MR-image (MP2RAGE).
Brain structure: Surface | Assessed at months 0 and 3
  Surface area (mm2) will be measured by a T1-weighted MR-image (MP2RAGE).
Brain structure: volumes of subcortical grey matter structures | Assessed at months 0 and 3
  Volumes (mm3) of subcortical grey matter structures will be measured by a T1-weighted MR-image (MP2RAGE).
Fasting concentration of peripheral blood mononuclear cells. | Assessed at months 0 and 3
  The concentration of isolated blood mononuclear cells will be measured in blood in fasting state.
Fasting concentration of sex hormones | Assessed at months 0 and 3
  The concentration of sex hormones will be measured in blood during fasting.
Puberty stage | Assessed at months 0, 3 and 9.
  Puberty stage will be evaluated by a standardized questionnaire completed by the parents that assesses the child's puberty stage according to the Tanner's stage classification method.

CONTACTS AND LOCATIONS:
Overall Officials: Faidon Magkos, PhD, Principal Investigator — University of Copenhagen, Department of Nutrition, Exercise and Sports
Locations (2):
- Denmark (2):
  - University of Copenhagen, Copenhagen
  - Faidon Magkos, Hvidovre

IPD SHARING:
Plan to Share IPD: No